CLINICAL TRIAL: NCT03081884
Title: Validation of FACBC as an Early Indicator of Sub-clinical Metastatic Disease Among High-risk Prostate Cancer Patients With Presumed Localized Disease
Brief Title: Validation of FACBC for Detection of Metastasis Among High-risk Prostate Cancer Patients With Presumed Localized Disease
Acronym: EDRN-FACBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David M Schuster, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00092595; U01CA113913-11 (NIH)
Record Dates: First submitted 2017-02-28; First posted 2017-03-16 (Actual); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Cancer
Keywords: Prostate cancer; Metastatic cancer; Urogenital disorders; Oncology; Radiology
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Neoplasm Metastasis; Urogenital Diseases | interventions — fluciclovine F-18

STUDY DESIGN:
Intervention Model Description: All participants will have the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FACBC PET-CT Imaging (Experimental): Individuals who have been diagnosed with primary prostate carcinoma and do not have definitive findings of systemic metastasis with conventional imaging will have a whole body FACBC PET-CT scan.
  Interventions: Drug: FACBC PET-CT Imaging

INTERVENTIONS:
Drug: FACBC PET-CT Imaging — Participants will fast for 4 hours to normalize their neutral amino acid levels. One hour prior to the scan, participants will drink up to 450ml of standard oral contrast. Participants will lie on the scanning bed while the bed moves through the PET/CT scanner for the CT portion of the exam. After completion of the CT scan, approximately 10 units of FACBC will be injected for the PET scan portion of the exam. The bed will move through the scanner again and the PET portion of the exam will take 30 minutes. The entire visit will take about two hours.
  Standard of care procedures include conventional imaging (CT and/or MRI; bone scan and/or NaF PET per institutional standards) and radical prostatectomy with extended pelvic lymph node dissection.
  Other Names: Fluciclovine

SUMMARY:
This study is for patients who have a high risk of metastatic prostate cancer (cancer that has spread outside of the prostate) who are going to have radical prostatectomy. The Anti-1-amino-3-[18F]fluorocyclobutyl-1-carboxylic acid (FACBC or Fluciclovine) positron emission tomography (PET) scan is a new imaging approach that has promising results in showing progression of cancer. The goal of this study is to determine if FACBC PET imaging will detect metastatic disease in patients with high risk prostate cancer who have negative conventional cross-sectional imaging such as computed tomography (CT) and/or magnetic resonance imaging (MRI), as well as bone scan and/or sodium fluoride PET. FACBC PET imaging may help detect metastatic prostate cancer in patients with newly diagnosed high risk primary prostate cancer and potentially improve staging of the cancer. Additionally, the researchers will compare the FACBC uptake in the prostate with uptake of FACBC detected in metastasis. They will also analyze and compare the prostate tissue, serum and urine parameters that are linked to higher rates of FACBC positivity.

DETAILED DESCRIPTION:
Approximately 50-80% of patients who are considered high-risk after being treated with definitive radical prostatectomy experience recurrent disease, often because of undetected extra-prostatic metastatic disease prior to treatment. There is increasing evidence that performing radical prostatectomy in patients with high-risk disease or locally advanced disease is feasible and has potential benefits in terms of local control, overall survival, and quality of life. Thus, improved imaging approaches for early detection of occult metastatic prostate cancer at the time of presentation could inform a directed treatment approach that would significantly improve patient outcomes, including use of extended lymphadenectomy as well as postoperative radiation therapy planning.

Amino acid transport is up-regulated in prostate and other cancers. Anti-1-amino-3-[18F]fluorocyclobutyl-1-carboxylic acid (FACBC) is a synthetic amino acid analog positron emission tomography (PET) radiotracer that has demonstrated promising results in the staging and restaging of prostate carcinoma, with high positive predictive value (PPV) in the identification of extraprostatic malignancy. Most of the prior studies of FACBC were in post-primary treatment recurrence, and this proposed trial will be the first comprehensive study to evaluate FACBC PET in detecting occult metastatic disease at initial diagnosis in patients with negative or equivocal conventional imaging, with the objective of developing a more effective primary treatment plan.

The goal of this study is to determine if FACBC PET will detect significant occult metastatic disease in patients with high risk primary prostate carcinoma who have negative or equivocal conventional imaging such as CT and/or MRI and bone scan. Participants will have a single scan prior to surgery for this study. Participants will be followed, through medical record reviews, for 10 years but no additional procedures related to this study will be performed.

ELIGIBILITY:
Inclusion Criteria:

* High-risk prostate cancer patients eligible for standard of care surgery

  * At least clinical T3a disease, and/or Gleason≥8, and/or Prostate-Specific Antigen (PSA) >20, as per clinical assessment and routine guidelines
* Undergone standard of care conventional imaging (CT and/or MRI; bone scan and/or sodium fluoride (NaF) PET)

Exclusion Criteria:

* Definitive findings of systemic metastasis on conventional imaging.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Alemozaffar, Principal Investigator — Emory University; David M Schuster, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alemozaffar M, Akintayo AA, Abiodun-Ojo OA, Patil D, Saeed F, Huang Y, Osunkoya AO, Goodman MM, Sanda M, Schuster DM. [18F]Fluciclovine Positron Emission Tomography/Computerized Tomography for Preoperative Staging in Patients with Intermediate to High Risk Primary Prostate Cancer. J Urol. 2020 Oct;204(4):734-740. doi: 10.1097/JU.0000000000001095. Epub 2020 Apr 29. PMID 32347780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began March 1, 2017 and all study follow-up was completed by December 31, 2019. Participants were enrolled from the patient population at Emory University Hospital in Atlanta, Georgia.
Groups:
- FACBC PET-CT Imaging: Individuals diagnosed with primary prostate carcinoma and without definitive findings of systemic metastasis with conventional imaging, had a whole body FACBC positron emission tomography (PET)-computerized tomography (CT)(PET-CT) scan followed by robotic radical prostatectomy with extended pelvic lymph node dissection.
Period: Overall Study
Arm/Group | FACBC PET-CT Imaging
Started | 61
Completed | 57
Not Completed | 4
Not completed — deferred prostate cancer treatment | 1
Not completed — metastasis managed with systemic therapy | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes participants who completed the study.
Arm/Group | FACBC PET-CT Imaging
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57
Type of Standard of Care Imaging [Count of Participants; unit: Participants]
  Computerized tomography (CT) | 20
  Magnetic resonance imaging (MRI) | 37

OUTCOME MEASURES:

1. Primary Outcome: Cancer Detection Performance of FACBC PET/CT
Description: The performance of FACBC PET/CT for diagnosing metastatic cancer was determined by confirming the FACBC PET/CT findings to the histological analysis of the lymph nodes.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- FACBC PET-CT Imaging: Individuals diagnosed with primary prostate carcinoma and without definitive findings of systemic metastasis with conventional imaging, had a whole body FACBC PET-CT scan followed by robotic radical prostatectomy with extended pelvic lymph node dissection.
Arm/Group | FACBC PET-CT Imaging
Number analyzed (Participants) | 57
Participants
  True positive | 17
  True negative | 22
  False positive | 4
  False negative | 14

2. Secondary Outcome: Diagnostic Performance of FACBC PET/CT and Conventional Imaging
Description: The diagnostic performance of FACBC PET/CT in the detection of extraprostatic disease is compared to the diagnostic performance of standard imaging, as confirmed with lymph node histology.
Time Frame: Day 1, Day of surgery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Conventional Imaging: Study participants also had conventional imaging (CT or MRI) as part of standard of care.
Arm/Group | FACBC PET-CT Imaging | Conventional Imaging
Number analyzed (Participants) | 57 | 57
percentage of participants
  Sensitivity | 55.3 [43.0 to 68.0] | 33.3 [21.0 to 47.0]
  Specificity | 84.8 [75.0 to 94.7] | 84.1 [73.3 to 94.4]
  Positive predictive value | 81.5 [69.2 to 93.3] | 72.2 [55.6 to 88.9]
  Negative predictive value | 60.8 [47.8 to 73.7] | 51.2 [40.0 to 63.0]
  Accuracy | 68.5 [59.4 to 78.1] | 56.3 [47.2 to 65.7]

ADVERSE EVENTS:
Time Frame: Adverse events were documented beginning at the time when the radiotracer was administered and ending 7 days after administration.
Arm/Group | FACBC PET-CT Imaging
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT03081884/Prot_SAP_000.pdf